CLINICAL TRIAL: NCT06316778
Title: Pelvic Floor Muscle Training for Urinary Incontinence in Women with Myotonic Dystrophy Type 1: a Feasibility and Acceptability Study
Brief Title: Pelvic Floor Muscle Training for Women with Myotonic Dystrophy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); Interdisciplinary research team on neuromuscular diseases (GRIMN) (Unknown); CIUSSS Saguenay-Lac-Saint-Jean (Unknown)
Responsible Party: Principal Investigator, Mélanie Morin, Researcher and full professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-038
Record Dates: First submitted 2024-03-07; First posted 2024-03-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Myotonic Dystrophy Type 1; Urinary Incontinence
Keywords: Neuromuscular disease; Physiotherapy; Exercises; Urinary incontinence
MeSH Terms: conditions — Myotonic Dystrophy; Urinary Incontinence; Neuromuscular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: pre-treatment assessment - intervention (12 weeks) - post-treatment assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pelvic floor muscle training (Experimental)
  Interventions: Behavioral: Pelvic floor muscle training

INTERVENTIONS:
Behavioral: Pelvic floor muscle training — 12 weekly sessions of 60 minutes with an experienced physiotherapist, including pelvic floor muscles (PFM) exercises with biofeedback, teaching home exercises and education.

SUMMARY:
Myotonic dystrophy type 1 (DM1) is a neuromuscular disease characterized by multisystem manifestations. DM1 can affect the urinary system through the impact of the pelvic floor muscles (PFM). Urinary incontinence can occur in this situation and is often offset with compensatory measures without restoring the PFM function (e.g. sanitary pads). PFM training have already been shown to be effective in reducing or even eliminating urinary incontinence in the general population. However, no study has been the subject of this modality in people with DM1. Having recently shown that it is possible to gain strength with DM1, a strengthening protocol targeting PFM could prove effective in treating urinary incontinence. The objectives of this study are i) to assess the feasibility and acceptability of PFM training and ii) to investigate the effects of PFM training in women with DM1 with adult phenotype. A quasi-experimental study will be conducted with 12 women having a confirmed diagnosis of DM1 with urinary incontinence. Participants will follow a 12-week PFM training program, comprising weekly sessions with an experienced physiotherapist as well as a home exercise program. Outcomes measures will be assessed at baseline and at post-treatment and will include: feasibility and acceptability variables, frequency of urinary incontinence, urogynecological symptoms and their impact on quality of life, morphometry and function of PFM, and the perceived improvement following the treatments. This study has the potential to improve the management of urinary incontinence and support the implementation of pelvic floor rehabilitation services in this population.

ELIGIBILITY:
Inclusion Criteria:

* confirmed medical diagnosis of myotonic dystrophy type 1 (DM1) with adult phenotype
* symptoms of stress, urge or mixed urinary incontinence
* able to give a free and informed consent

Exclusion Criteria:

* being pregnant, have given birth by vaginal delivery in the last year or plan to become pregnant in the next six months
* present post-void residual urine ≥ 150 ml
* have medical conditions that may have an impact on the symptoms of urinary incontinence and the response to treatments
* present fecal incontinence (≥ 1/week) or significant prolapse (beyond the hymen)
* have already received physiotherapy treatments in pelvic floor rehabilitation or surgery on the perineum
* have a defibrillator, pacemaker or bladder stimulator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of attended treatment sessions | Through treatment completion (session 1 to 12; 12 weeks of treatment)
  To determine feasibility, the patients' adherence to treatment sessions will be recorded (present vs absent) as well as reasons for non-attendance.
Percentage of home exercises performed | Through treatment completion (session 1 to 12; 12 weeks of treatment)
  1. The adherence rate to home exercises for each treatment group will be assessed using a daily diary. The participants will record the frequency of the exercises completed.
  2. To determine feasibility by assessing adherence to treatment sessions.
Retention rate | Baseline to Post-treatment assessment (2-week post-treatment)
  To determine feasibility by assessing the percentage of participants completing the post-treatment assessment. Reason for dropouts will be compiled.
Recruitment rate | Baseline
  To determine feasibility by assessing the percentage of participants included versus the participants screened. The barriers and reasons for refusing to participate as well as the reasons for exclusion will be documented.
Intervention Acceptability Questionnaire | At baseline and after 12 weeks of treatment
  The Intervention Acceptability Questionnaire will be used to assess the participants' acceptability of the interventions. This questionnaire consists of 4 items measured on a VAS scale (Minimum value: 0; Maximum Value: 10). Each item is analyzed separately, with a greater score meaning higher acceptability of the intervention. This outcome measure will contribute to identifying factors limiting the acceptability of each program.

SECONDARY OUTCOMES:
Change in the frequency of urinary incontinence episodes | Baseline to post-treatment (after the 12-week program)
  Evaluated with the 7-day bladder diary (number of leak/week).
Change in urinary incontinence symptoms | Baseline to post-treatment (after the 12-week program)
  Evaluated with the International Consultation Incontinence Questionnaire (ICIQ-UI-SF) Ranging from 0 to 21, higher scores indicate worse outcome (more urinary incontinence symptoms and a higher impact on their quality of life).
Change in pelvic floor disorder symptoms | Baseline to post-treatment (after the 12-week program)
  Evaluated with the Pelvic Floor Disorder Inventory (PFDI). Ranging from 0 to 300, higher scores indicate worse outcome (more pelvic floor disorder symptoms).
Change in pelvic floor disorder symptoms related impact on quality of life | Baseline to post-treatment (after the 12-week program)
  Evaluated with the Pelvic Floor Impact Questionnaire (PFIQ-SF). Ranging from 0 to 300, higher scores indicate a worse outcome (higher impact on their quality of life).
Change in pelvic floor muscles morphometry | Baseline to post-treatment (after the 12-week program)
  Evaluated with transperineal ultrasound.
Change in pelvic floor muscles function | Baseline to post-treatment (after the 12-week program)
  Evaluated with dynamometry.
Patient's satisfaction | Post-treatment (after the 12-week program)
  Evaluated with Patient satisfaction questionnaire (PSQ) ranging from "completely satisfied" to "not satisfied at all".
Patient's global impression of change | Post-treatment (after the 12-week program)
  Evaluated with Patients' Global Impression of Improvement (PGI-I). Ranging from 1 "very much better" to 7 "very much worse" on a 7-point likert scale.
Patient's estimated improvement | Post-treatment (after the 12-week program)
  Evaluated with Estimated percent improvement (EPI). Ranging from 0 "no amelioration" to 100 "complete amelioration".

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique des maladies neuromusculaires, Jonquière, Quebec, Canada